CLINICAL TRIAL: NCT06590077
Title: A Pilot Study to Investigate the Impact of Aromatherapy on Wellbeing and Relaxation in Gynae Oncology Patients Post Treatment
Brief Title: Impact of Aromatherapy on Wellbeing and Relaxation in Gynae Oncology Patients Post Treatment
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Dublin, Trinity College (Other)
Collaborators: St. James's Hospital, Ireland (Other)
Responsible Party: Principal Investigator, Astrid Sasse, Associate Professor, University of Dublin, Trinity College
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 4308-24072024
Record Dates: First submitted 2024-09-06; First posted 2024-09-19 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Stress; Wellbeing; Relaxation
Keywords: Aromatherapy; Inhalation; Essential Oil; Complementary Therapy; Stress and anxiety; Relaxation and wellbeing
MeSH Terms: conditions — Respiratory Aspiration; Anxiety Disorders | interventions — Aromatherapy; Oils, Volatile; Population Groups

STUDY DESIGN:
Intervention Model Description: A double-blind, randomised controlled experiential pilot study with a test and a control product both of which contain essential oil fragrances.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Test blend of five essential oils in a carrier oil - rollerball (Active Comparator): The test product contains a blend of 5 essential oils (orange, lavender, frankincense, vetiver, and neroli), diluted in apricot kernel oil. It was formulated by a clinical aromatherapist (Fiona Hedigan) to promote wellbeing and aid relaxation. To date there have been no reports of adverse events. Permission has been given to supply this formula for the research study. The rollerball product ('REST') is available commercially under the FLORA & FIONA brand.
  Interventions: Other: Aromatherapy
- Control oil - rollerball (Placebo Comparator): Juniper essential oil in apricot kernel oil - presentation as a rollerball. The control oil has a mild aroma and is at low concentration.
  Interventions: Other: Control (placebo) group

INTERVENTIONS:
Other: Aromatherapy — The test intervention is an aromatherapy cosmetic product containing a blend of 5 essential oils (orange, lavender, frankincense, vetiver, and neroli), diluted in apricot kernel oil. It was formulated by a clinical aromatherapist. Each participant will be asked to use the product every evening over 4 weeks and to complete a validated questionnaire at 3 time points: at the beginning, midway after 2 weeks and at the end of the 4-week study.
  Other Names: Essential Oil; Aromatherapy Inhaler; Aromatherapy blend
  Arms: Test blend of five essential oils in a carrier oil - rollerball
Other: Control (placebo) group — Juniper essential oil in apricot kernel oil in low concentration with a faint aroma - presentation as a rollerball. Each participant will be asked to use the product every evening over 4 weeks and to complete a validated questionnaire at 3 time points: at the beginning, midway after 2 weeks and at the end of the 4-week study.
  Other Names: Essential oil - control
  Arms: Control oil - rollerball

SUMMARY:
The goal of this pilot study is to learn if aromatherapy helps to reduce stress and improve relaxation and wellbeing in gynaecological cancer patients after they have finished their treatment for cancer. The main questions this study aims to answer are:

Is there a benefit in using an aromatherapy product for relaxation and wellbeing after completion of cancer treatment.

Researchers will compare a commercially available aromatherapy test oil blend to a control oil (an oil at high dilution with a faint aroma) to see if the oil blend helps to reduce stress and increase wellbeing and relaxation.

Participants will:

Use a commercially available aromatherapy product or a control every evening for 4 weeks and complete a questionnaire at the start, after 2 weeks and at the end of the 4 week period.

During the four weeks of the study, the participants may wish to record their experience with the test oil and assess its impact on relaxation and wellbeing in a personal diary.

DETAILED DESCRIPTION:
Patients will be identified by Prof Catherine O'Gorman who directs the Gynae-oncology survivorship clinic. Patients who attend the clinic are at least 6 months post treatment for their gynaecological cancer. Patients wo are referred to the clinic undergo a holistic needs assessment as part of their care at the clinic. Following completion of the assessment, Prof O'Gorman will identify patients who would be eligible for the study and supply them with the patient information leaflet and consent form. Those who wish to participate will be contacted by the researcher (Fiona Hedigan) to arrange a meeting in St. James's Hospital.

Patients who have been identified as eligible for the study by Prof O'Gorman will receive a patient information leaflet and consent form at their clinic visit. Those who express an interest in participating in the study will be contacted by the researcher (Fiona Hedigan) who will arrange to meet the patient on site in St. James's Hospital. During the meeting, the study will be explained in detail and the researcher will go through the patient information leaflet and consent form with the patient. If the patient agrees to participate, the consent form will be completed in person with the patient and a copy of the signed consent given to the patient for their records.

Participants will be asked to use an aromatherapy cosmetic product every evening for four weeks and assess its impact on relaxation and wellbeing. The participants will be asked to complete a questionnaire three times: at the start of the study, midway after 2 weeks, and at the end of the 4th week. The test intervention is an aromatherapy cosmetic product containing a blend of 5 essential oils (orange, lavender, frankincense, vetiver, and neroli), diluted in apricot kernel oil. It was formulated by the postgraduate researcher who is a clinical aromatherapist. To date there have been no reports of adverse events. Permission has been given to supply this formula for the research study. The control product will contain a single essential oil (juniper) with a mild aroma at a low concentration diluted in apricot kernel oil.

The Warwick, Edinburgh Mental Wellbeing Scale (WEMWBS) is a validated and effective tool used to measure levels of wellbeing. Initial feedback from using the product will also be obtained by completion of an organoleptic profile survey.

Data from all 3 questionnaires will be pseudonymous, however all the questionnaires responses can be linked via the ID number on the aromatherapy product which participants will insert when completing each survey.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are 6 months post active treatment attending the gynae oncology clinic at St James's Hospital, Dublin, Ireland.
* Adult with capacity to provide informed consent

Exclusion Criteria:

* Anyone who has a hypersensitive reaction to aromatic fragrances.
* Pregnant or planning a pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-08-19 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Primary outcome: To measure the effect of an aromatherapy cosmetic product on the levels of relaxation and wellbeing in the participants as determined by questionnaire after four weeks | 4 weeks
  Each participant will complete a validated questionnaire at 3 time points: at the beginning, midway after 2 weeks and at the end of the 4-week study.
  The Warwick, Edinburgh Mental Wellbeing Scale (WEMWBS) is a validated and effective tool used to measure levels of wellbeing. Wellbeing scores range from 14 (poor wellbeing) to 70 where 70 is 'high wellbeing'.
  Data from all 3 questionnaires can be linked via the ID number on the aromatherapy product which participants will insert when completing each survey.
  The primary outcome measure will compare the questionnaire at the beginning of the study with the questionnaire at the end of the four week period.

SECONDARY OUTCOMES:
Focus Group after completion of the 4 week study | October to December 2024
  Conduct in-person focus groups on site in the hospital to gain further feedback of using the aromatherapy rollerball product.
To measure the effect of an aromatherapy cosmetic product on the levels of relaxation and wellbeing in the participants as determined by questionnaire after two weeks | 2 weeks
  Each participant will complete a validated questionnaire at 3 time points: at the beginning, midway after 2 weeks and at the end of the 4-week study.
  The Warwick, Edinburgh Mental Wellbeing Scale (WEMWBS) is a validated and effective tool used to measure levels of wellbeing. Wellbeing scores range from 14 (poor wellbeing) to 70 where 70 is 'high wellbeing'.
  Data from all 3 questionnaires can be linked via the ID number on the aromatherapy product which participants will insert when completing each survey.
  The secondary outcome measure will compare the questionnaire at the beginning of the study with the questionnaire at the end of the two week period.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine O Gorman, MD, Principal Investigator — St. James Hospital, Dublin, Ireland; Astrid Sasse, Principal Investigator — University of Dublin, Trinity College
Locations (1):
- St. James Hospital, Dublin, Ireland, Dublin, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: No
This was not part of our ethics application.